CLINICAL TRIAL: NCT05818436
Title: Impact on General Functionality of an Immediate Prosthetic Functionalization Protocol in People Over 70 Years of Age with Deficient Removable Prostheses
Brief Title: Immediate Dental Prosthesis Functionalization Protocol in People Over 70 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: National Fund for Research and Development in Health, Chile (Other)
Responsible Party: Principal Investigator, Pilar Barahona, Principal Investigator, Clinical Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05595304
Record Dates: First submitted 2023-03-08; First posted 2023-04-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Dental Prosthesis Failure; Frail Elderly Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Oral Functionalization Prosthesis repairment (Experimental): Experimental: Oral Functionalization Prosthesis repairment: prosthetic reline and occlusal stabilization through repair of missing pieces and recovery of occlusal contacts and follow up with conventional prosthesis treatment
  Interventions: Procedure: Procedure: prosthetic functioning; Device: Conventional dental prosthesis
- Active Comparator: control (Active Comparator): Active Comparator: control conventional prosthetic treatment (new prosthesis)
  Interventions: Device: Conventional dental prosthesis

INTERVENTIONS:
Procedure: Procedure: prosthetic functioning — Prosthetic reline and occlusal stabilization through repair of missing pieces and recovery of occlusal contacts
  Arms: Experimental: Oral Functionalization Prosthesis repairment
Device: Conventional dental prosthesis — : conventional prosthetic treatment new prosthesis

SUMMARY:
Sarcopenia and malnutrition are closely involved in frailty. To prevent them, it is essential to assess oral function. "Oral fragility" manifests with specific signs or symptoms, including occlusion loss due to tooth loss and chewing difficulty. To recover from it, restoring function by placing a dental prosthesis in the event of tooth loss is essential. In Chile, many patients referred to secondary care to perform new prosthetic treatment live in conditions of less oral functionality and enter waiting lists that can take years, impacting general functionality. Falls are a public health problem with a high economic cost, the second cause of death worldwide. One of the causes is sarcopenia, and it has been studied that the decrease in the number of teeth and the occlusal posterior support region may be risk factors for decreased gait speed, an objective measurement of fall risk. It has been studied that the decrease in the number of teeth causes a reduction in total muscle mass, walking speed and lower quality of life.

General objective: To evaluate the impact on the general functionality of applying an immediate prosthetic functionalization protocol in patients with deficient removable prostheses, compared with conventional treatment, at the secondary level of the health system, in patients over 70 years of age.

Methodology: randomized, double-blind clinical trial with two groups of 62 patients each: experimental and control. The intervention will consist of recovering prosthetic function in one session before conventional rehabilitation vs the control group receiving conventional rehabilitation. Measurements will include manual grip strength measurements made with a Jamar dynamometer, timed up-and-go test, before and after prosthetic treatments and quality of life related to oral health through Ohip 7sp. Descriptive statistics will be applied through the registration of frequency and contingency tables. To compare hand grip strength, Pearson's Correlation will be used; for risk of pre and post-fall, the t-test will be applied for two related samples; for quality of life before and after the intervention, Chi2 will be used; changes in grip strength, fall risk and quality of life, between the different groups according to the Eichner index, one-way ANOVA will be applied, for related samples.

DETAILED DESCRIPTION:
In the public health system, older adults who need new dental prostheses are referred from primary health care to the rehabilitation speciality at the secondary care level. In many cases, they wear old, fractured, non-functional prosthetic devices and enter waiting lists for several months at the hospital level. During that time, they continue a process of oral hypofunction, which gradually progresses to a process of oral dysfunction and decreased systemic function. Once they are called from the secondary level to enter treatment, they must wait for the rehabilitation process, which takes about two months, a period in which they continue with oral hypofunction. This functional pathophysiological condition closely maintains the negative impact on nutrition. Our proposal consists of carrying out a dental intervention, the competence of the general dentist when the patient begins the conventional treatment process, once you enter secondary care. This intervention is intended to immediately recover bilateral, homogeneous and simultaneous occlusal contacts and recover the prosthetic biomechanical characteristics by improving prosthetic support, retention and stability. This will be made with supplies commonly used in the dental clinic, health services and university teaching clinics. To evaluate this intervention's effect at the muscular level, the patient's manual grip strength and gait speed will be measured before the intervention and fifteen days later. Subsequently, once the new prostheses have been made, a new measurement will be made. Quality of life survey related to oral health will be applied to both groups before and after the intervention and treatment. Based on international scientific evidence and on an investigation carried out by this research team (presented at the Chilean National Congress of Geriatrics and Gerontology), between October 2018 and April 2019 in 60 octogenarian older adults not wearing prostheses in whom dental prostheses were built - whose objective was to determine if there was an association between the use of prostheses that return the premolars and molars and the gripping force of the hand. Hand tightening force was measured before and 15 days after prosthetic rehabilitation with a manual hydraulic dynamometer (Jamar MR). For the cohort in the study, the use of prostheses increased the hand's gripping force by a statistically significant value.

This research aims to contribute to the Chilean population since the immediate recovery of oral functionality may contribute to reducing conditions that increase frailty, which in cases of entering long-term lists is expected to have a more significant impact on the systemic level and higher health costs.

In some cases, out-of-pocket spending on dental supplies will also be reduced because by recovering prosthetic biomechanical conditions, older people will not have to invest resources in creams and adhesive powders to "improve" prosthetic adhesion. With this, it is also possible to contribute to improving the quality of life of these patients due to the recovery of functions: masticatory and social. It will also allow better integration of dentists into the multidisciplinary team in the care model proposed by the Health Ministry. It will allow the development and implementation of a care protocol in primary health care, considering that the intervention will contemplate actions that are the responsibility of general dentists.

Without the development of this research, the care system will maintain its long waits for this age group for treatment, a situation that will continue to increase considering that global projections related to a greater increase in older inhabitants and also the costs already described

ELIGIBILITY:
Inclusion Criteria:

* 70 or older
* Willingness to participate
* Discharged from Primary Care to the Oral Health Department at Hospital Salvador, Santiago Chile for prosthetic treatment
* With both maxilar an mandibular prosthesis affected
* Eichner groups B3, B4, C1, C2 and C3.

Exclusion Criteria:

* Cognitive impairment (Pfeiffer test classified as moderate or severe)
* Diseases that affect the ability to use facial muscles
* Soft Tissue diseases that affect facial functionality like fibroids

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Handgrip strength change | Time Frame: Baseline, 15 and 30 days after intervention
  measurment in kilograms of handgrip strength. Higher scores mean a better outcome
Time up-and-go change | Time Frame: Baseline, 15 and 30 days after intervention
  Measurement of Timed up-and-go test. Measured in seconds. Higher scores mean worse outcomes
Estimation of oral health-related Quality of Life change | Time Frame: Baseline, 15 and 30 days after intervention
  Use of Oral Health Impact Profile Ultra Short Version (OHIP 7Tsp) survey. Score from 0 to 28, higher scores mean worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Pilar O Barahona, DDS, MSC, Study Chair — University of Chile
Locations (1):
- Hospital Salvador, Santiago, Santiago Metropolitan, Chile